CLINICAL TRIAL: NCT01161576
Title: Direct CNS Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Serotype rh.10 Expressing the Human CLN2 cDNA to Children With Late Infantile Neuronal Ceroid Lipofuscinosis (LINCL)
Brief Title: Safety Study of a Gene Transfer Vector (Rh.10) for Children With Late Infantile Neuronal Ceroid Lipofuscinosis (LINCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0810010013; UL1TR000457-06 (NIH)
Record Dates: First submitted 2010-03-22; First posted 2010-07-13 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Batten Disease; Late-Infantile Neuronal Ceroid Lipofuscinosis
Keywords: Batten Disease; Late Infantile Neuronal Lipofuscinosis; gene transfer
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Intervention Model Description: We chose an initial dose two fold lower of 9.0x10^11 genome copies/subject (Group A). Initially, the study plan was to proceed to Group B, which would receive a higher dose of 1.8x10^12 genome copies if the initial dose was well tolerated. However, after assessing the MRI images of the first 6 children who received the dose of 9.0x10^11 gc, we discovered that 4 of the 6 subjects at 6 months and 1 of the 6 subjects at 12 months exhibited varying degrees of T2 hyperintensities related to diffusion restriction at the sites of vector deposition. Although there are no clinical correlates to these MRI findings, we have decided to lower the dose by ½ log to 2.85x10^11 gc for the remaining subjects to be enrolled in protocol #0810010013. The volume of the drug solution will be the same as in Group A, but the concentration of the vector will be ½ log less.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The first dose cohort consists of 6 subjects who received AAVrh.10CUhCLN2 vector 9.0x10^11 genome copies (gc) total dose. This is equal to 900,000,000,000 molecules of the drug.
  Interventions: Biological: AAVrh.10CUhCLN2 vector 9.0x10^11 genome copies
- Group B (Experimental): The second dose cohort consists of 10 subjects, who will receive AAVrh.10CUhCLN2 vector 2.85x10^11 genome copies (gc) total dose. This is equal to 285,000,000,000 molecules of the drug.
  Interventions: Biological: AAVrh.10CUhCLN2 vector 2.85x10^11 genome copies

INTERVENTIONS:
Biological: AAVrh.10CUhCLN2 vector 9.0x10^11 genome copies — The experimental drug for this second generation study has a genome identical to that used in our previous study and delivers the same gene, but instead of an AAV2 capsid (protein shell of the virus), the new vector has the capsid of AAVrh.10, a clade E AAV derived from rhesus macaque (a species of Old World monkeys). The first dose that was given to the first 6 subjects is 9.0x10^11(900,000,000,000 molecules of the drug) genome copies/subject. In regards to drug administrations, we propose to perform 2 series of 6 simultaneous administrations of vector for 75 min each. Each subject will receive the assigned dose of AAVrh.10CUhCLN2, divided among 12 locations delivered through 6 burr holes (2 locations at 2 depths through each hole), 3 burr holes per hemisphere.
  Arms: Group A
Biological: AAVrh.10CUhCLN2 vector 2.85x10^11 genome copies — The experimental drug for this 2nd generation study has a genome identical to that used in our previous study and delivers the same gene but instead of an AAV2 capsid (protein shell of the virus), the new vector has the capsid of AAVrh.10, a clade E AAV derived from rhesus macaque (a species of Old World monkeys). Group B will receive a dose of 2.85x10^11 genome copies (285,000,000,000 molecules of the drug). In regards to drug administration, we propose to perform 2 series of 6 simultaneous administrations of vector for 75 min each. Each subject will receive the assigned dose of AAVrh.10CUhCLN2, divided among 12 locations delivered through 6 burr holes, 3 burr holes per hemisphere.
  Arms: Group B

SUMMARY:
This is a proposed follow up study on the investigators previous gene transfer human clinical trial entitled "Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Expressing the Human CLN2 cDNA to the Brain of Children with Late Infantile Neuronal Ceroid Lipofuscinosis" (Weill Cornell IRB# 0401007010). As in the previous study, the investigators propose to administer a biologic by direct gene transfer into the brain and assess its safety on children with a fatal genetic disease of the central nervous system (CNS). The disease is Late Infantile Neuronal Ceroid Lipofuscinosis (LINCL, a form of Batten disease). This will be accomplished by using delivery of a gene (method called gene transfer) to administer to the brain an experimental drug called AAVRh.10CUhCLN2, a gene transfer vector.

DETAILED DESCRIPTION:
The investigators propose to assess a new drug to treat children with a form of Batten Disease called Late Infantile Neuronal Ceroid Lipofuscinosis (LINCL). These children are born with genetic changes called mutations in their CLN2 gene that result in the inability of the brain to properly recycle proteins. The recycling failure leads to death of the nerve cells in the brain and progressive loss of brain function. Children with Batten disease are normal at birth but by age 2 to 4 have motor and vision problems which progress rapidly to death at age approximately 10 years old. There are no therapies available to treat the disease.

The experimental gene transfer procedure treatment the investigators propose consists of augmenting the abnormal gene by a good copy. A virus is used to deliver the good gene to the nerve cells. Since the disease is due to an abnormal CLN2 gene, the aim of this study is to add a normal copy of the CLN2 gene to the brain of affected children to try to reverse death of cells in the brain. Previously the investigators have used a virus called adeno-associated virus 2 (AAV2) as the gene delivery system. That study showed that viral delivery of the gene was safe. We now propose to use a slightly different virus called AAVrh.10 as a gene delivery system and use 2 different doses of the virus. Children with Batten disease will get the drug injected into the brain and will receive extensive neurological assessment at intervals to determine if the transfer slows the rate of progress of the disease.

The primary aims of the study are: (1) to assess the hypothesis that direct administration of AAVrh.10CUhCLN2 to the brain of children with LINCL can be achieved safely and with minimal toxicity; and (2) to evaluate the hypothesis that direct administration of AAVrh.10CUhCLN2 to the brain of children with LINCL will slow down or halt progression of the disease as assessed by neurological rating scales and quantitative MRI (primary variables).

The investigators have recently completed a study in which the normal copy of the gene was surgically delivered to 12 locations in the brain in 10 children with LINCL. The children were assessed by a number of neurological and imaging parameters prior to and after gene transfer. The data demonstrated that the gene transfer was well tolerated and had a small impact on the progression of the disease and suggested that higher doses and a better delivery system may provide greater benefit. The previous study used the viral gene transfer vector adeno-associated virus type 2 (AAV2) at a dose of 2,000,000,000,000 molecules of the drug (2 x 10^12 particle units). The investigators now propose a very similar study with delivery of the identical payload with a slightly different viral gene delivery system based on the virus AAVrh.10.

ELIGIBILITY:
Inclusion Criteria:

All individuals who meet the following criteria will be included without bias as to a gender or race/ethnicity. Each case will be individually reviewed with the Eligibility Committee comprised of 3 physicians other than the PI, including a pediatric neurosurgeon, pediatric neurologist and general pediatrician.

1. Definitive diagnosis of LINCL, based on clinical phenotype and genotype. The genotype must include at least one of the 5 most common CLN2 mutant genotypes: C3670T (nonsense Arg208 to stop), G3556C (intron 7 splice), G5271C (Gln422His), T4396G (aberrant splicing, intron 8) and G4655A (Cys365Tyr). If either parental allele is R447H, the patient will not be included in the study. These account for a total of 83% of the mutations in the study by Sleat et al and 82% of the mutations in our studies. The study does not limit to one specific genotype (genetic constitution) since our data regarding the natural history of the disease and the studies of Steinfeld, show that, for these 5 genotypes (genetic constitution), LINCL subjects have similar clinical course.
2. The subject must be between the age of 2 and 18 years.
3. Subjects will have an average total score of 4 - 12 on the Weill-Cornell LINCL scale, and the total score should not be outside the 95th percentile confidence limits for age based on our historic data.
4. The subject will not previously have participated in a gene transfer or stem cell study.
5. Parents of study participants must agree to comply in good faith with the conditions of the study, including attending all of the required baseline and follow-up assessments, and both parents or legal guardians must give consent for their child's participation.
6. Sexually active subjects will have to use contraception during the treatment and for 2 months after completion of the treatment.
7. If asymptomatic (i.e - An LINCL score of 12), has one older sibling who has a positive genotype and has clinical manifestations of the disease.

Exclusion Criteria:

1. Presence of other significant medical or neurological conditions may disqualify the subject from participation in this study, particularly those which would create an unacceptable operative risk or risk to receiving the AAVrh.10CUhCLN2 vector, e.g., malignancy, congenital heart disease, liver or renal failure.
2. Subjects without adequate control of seizures.
3. Subjects with heart disease that would be a risk for anesthesia or a history of major risk factors for hemorrhage.
4. Subjects who cannot participate in MRI studies.
5. Concurrent participation in any other FDA approved Investigational New Drug.
6. Subjects with history of prolonged bleeding or abnormal platelet function or taking aspirin.
7. Renal disease or altered renal function as defined by serum creatinine > 1.5 mg/dl at admission.
8. Abnormal serum sodium, potassium calcium, magnesium, phosphate at grade III or IV by Division of AIDS Toxicity Scale.
9. Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and or Total Bilirubin > 1.3 mg/dL
10. Immunosuppression as defined by WBC < 3,000/µL at admission
11. Uncorrected coagulopathy during the baseline period defined as INR > 1.4; PTT > 35 sec; PLT < 100,000/mm3.
12. Anemia (hemoglobin < 11.0 g/dl at > 2 years of age, with normal serum iron studies).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08-19 (Actual); Primary Completion 2016-01-05 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Weill-Cornell LINCL scale from Baseline to 18 months | 18 Months
  A clinical rating, 12 point scale which combines assessment of feeding, gait, motor and language to give an overall assessment of various CNS functions.
Disease progression based on change in MRI imaging parameter (% grey matter volume) from Baseline to 18 Months | 18 Months
  Based on previous analyses, we have determined that 3 imaging parameters (% grey matter volume, MRI Assessment, % ventricular volume and cortical apparent diffusion coefficient) correlate best with age and with the Weill Cornell LINCL scale and will be used to assess disease progression and the effect of the gene transfer.
Disease progression based on change in MRI imaging parameter (% ventricular volume) from Baseline to 18 Months | 18 Months
  Based on previous analyses, we have determined that 3 imaging parameters (% grey matter volume, MRI Assessment, % ventricular volume and cortical apparent diffusion coefficient) correlate best with age and with the Weill Cornell LINCL scale and will be used to assess disease progression and the effect of the gene transfer.
Disease progression based on change in MRI imaging parameter cortical apparent diffusion coefficient) from Baseline to 18 Months | 18 Months
  Based on previous analyses, we have determined that 3 imaging parameters (% grey matter volume, MRI Assessment, % ventricular volume and cortical apparent diffusion coefficient) correlate best with age and with the Weill Cornell LINCL scale and will be used to assess disease progression and the effect of the gene transfer.

SECONDARY OUTCOMES:
Change in Quality of Life Survey from Baseline to 18 Months | 18 months
  The quality of life survey that will be completed by at least one parent/legal guardian at the screening visit and the month 18 visit will be either the Infant Toddler Quality of Life (ITQoL) questionnaire or the Child Health Questionnaire (CHQ), depending on the age of the subject. The ITQoL is administered to subjects up to the age of five and the CHQ is administered to subjects from age 5-18.
Mullen Scale (developmental assessment) from Baseline to 18 Months | 18 months
  Averaging the scores from the Mullen Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De BP, Cram S, Lee H, Rosenberg JB, Sondhi D, Crystal RG, Kaminsky SM. Assessment of Residual Full-Length SV40 Large T Antigen in Clinical-Grade Adeno-Associated Virus Vectors Produced in 293T Cells. Hum Gene Ther. 2023 Aug;34(15-16):697-704. doi: 10.1089/hum.2023.032. PMID 37171121